CLINICAL TRIAL: NCT01498614
Title: Psychological Impact, Metabolic Control, and Biological Stress Markers in Diabetes: Intervention Study With Affect School and Basal Body Awareness
Brief Title: Psychological Impact in Diabetes: Intervention With Affect School and Basal Body Awareness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator no longer at LU.
Sponsor: Lund University (Other)
Collaborators: Landstinget Kronoberg, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoU-Kronoberg Sweden 4522
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus; Depression; Alexithymia; Anxiety
Keywords: Diabetes mellitus; depression; anxiety; negative self image; alexithymia; metabolic control; diabetes complications
MeSH Terms: conditions — Diabetes Mellitus; Depression; Affective Symptoms; Anxiety Disorders; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Affect school (Experimental): Affect school is an educational intervention which includes 8 group sessions followed by 10 individual meetings with therapist
  Interventions: Behavioral: Affect School and Basal body awareness
- Basal body awareness (Active Comparator): Basal body awareness is an educational method with 9 group sessions followed by 6 individual meetings
  Interventions: Behavioral: Affect School and Basal body awareness

INTERVENTIONS:
Behavioral: Affect School and Basal body awareness — Affect School is an educational method based on SS Tomkins affect theory and Basal Body Awareness therapy is an educational stress reducing method

SUMMARY:
Psychological Impact, Metabolic Control, and Biological Stress Markers in Diabetes: Intervention Study With Affect School and Basal Body Awareness

Background:

Depression is common in patients with diabetes and is associated with impaired metabolic control. Alexithymia has been associated with depression, anxiety, stress related disorders and diabetes mellitus. Affect School (AS) is an intervention that may reduce depression and alexithymia according to previous research. Basic Body Awareness Therapy (BBA) is a stress-reducing technique.

Purpose:

Our aim is to: 1. Analyze the prevalence of depression and anxiety and the personality variables alexithymia and self image in diabetes patients. 2. Explore correlations between these variables and risk factors, including biochemical markers for diabetic complications. 3. To evaluate an intervention with AS and BBA in patients with diabetes that scored high in psychometric self-report tests and at the same time showed impaired metabolic control.

Method:

A randomized controlled trial of 350 people with diabetes, 18-59 years, 56% men, 44% women. Base-line study: from medical records and the National Diabetes Registry - waist circumference, BMI, blood pressure, type and duration of diabetes, diabetes complications, other diseases, medications, exercise habits and smoking. Tests - A1c, blood lipids, cytokines, hormones, beta-cell antibodies, c-peptide, midnight cortisol (salivary). Self-report tests of psychological and personality variables: HAD, TAS-20, SASB. Intervention: patients with A1c ≥ 8 and anxiety (HAD ≥ 8), depression (HAD ≥ 8), negative self-image (SASB: AFF <284) or alexithymia (TAS-20 ≥ 61) were randomized to AS or BBA. AS: 8 group sessions followed by 10 individual sessions. Instructors were a primary care physician and a psychotherapist. BBA: 9 group meetings and 6 individual sessions with a physiotherapist as instructor. Post intervention: Self report tests, A1c, cytokines, hormones, cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and type 2 diabetes at a specialist outpatient clinic in Vaxjo

Exclusion Criteria:

* Other severe somatic disorder, including being deaf or blind.
* Severe psychiatric disorder requiring psychiatric specialist care;
* psychotic disorder,
* bipolar disorder,
* severe drug abuse.
* Inadequate knowledge of Swedish.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 2009-03; Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression | 3 years
  Evaluate depression score before and after intervention

SECONDARY OUTCOMES:
Level of A1C | 3 years
  Compare the A1C level before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eva O Melin, MD, Principal Investigator — Landstinget Kronoberg, Sweden
Locations (1):
- Landstinget Kronoberg, Vaxjo, Kronoberg County, Sweden